CLINICAL TRIAL: NCT06461390
Title: The Effect of Fluid Loading With Early Norepinephrine Administration on Stroke Volume Index, Cardiac Index, Lactate, and Arterial Elastance in Pediatric Septic Shock
Brief Title: The Effect of Early Norepinephrine on Stroke Volume Index, Cardiac Index, Lactate, and Arterial Elastance in Pediatric Septic Shock
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Mulyono, Pediatrician, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-12-2106
Record Dates: First submitted 2024-06-04; First posted 2024-06-17 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Septic Shock; Sepsis
Keywords: pediatric septic shock; pulmonary edema; early norepinephrine; fluid loading
MeSH Terms: conditions — Shock, Septic; Sepsis; Pulmonary Edema | interventions — Norepinephrine; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: Interventional subject will be received fluid loading with early norepinephrine administration with dose 0.1 mcg/kgBW/minute control subject will be received fluid loading only
Masking Description: fluid loading with norepinephrie
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Norepinephrine Group (Fluid loading with early norepinephrine administration group) (Experimental): NE Group will receive ringer lactate bolus 20 ml/kg along with norepinephrine infusion at 0.1 mcg/kg/ minute until MAP>5 percentile.
  Additional fluid boluses of 10-20 ml/kg will be administered (up to a total of 60 ml/kg) until shock resolution or signs of fluid overload are observed, with or without continued norepinephrine infusion according to the treatment group
  Interventions: Drug: Norepinephrine
- Ringer's lactate Group (Active Comparator): The Fluid Group will receive only ringer lactate bolus 20 ml/kg. Additional fluid boluses of 10-20 ml/kg will be administered (up to a total of 60 ml/kg) until shock resolution or signs of fluid overload are observed.
  Interventions: Drug: Ringer's Lactate

INTERVENTIONS:
Drug: Norepinephrine — NE Group (Fluid loading with early norepinephrine administration group) NE Group will receive ringer lactate bolus 20 ml/kg along with norepinephrine infusion at 0.1 mcg/kg/minute until MAP>5 percentile. Additional fluid boluses of 10-20 ml/kg will be administered (up to a total of 60 ml/kg) until shock resolution or signs of fluid overload are observed, with or without continued norepinephrine infusion according to the treatment group
  Arms: Norepinephrine Group (Fluid loading with early norepinephrine administration group)
Drug: Ringer's Lactate — Fluid Group will receive ringer lactate bolus 20 ml/ kg only. Additional fluid boluses of 10-20 ml/kg will be administered (up to a total of 60 ml/kg) until shock resolution or signs of fluid overload are observed
  Arms: Ringer's lactate Group

SUMMARY:
The complexity of pediatric septic shock arise from its varied pathophysiology, which includes systemic inflammation, cardiovascular collapse, and multiple organ dysfunction. Current standard treatments, which primarily focusedon fluid resuscitation, had exhibited several problems. Excessive fluid resuscitation has been associated with complications such as fluid overload, which may cause conditions such as pulmonary edema and organ dysfunction, leading to worsened outcomes. This emphasizes the need for alternative therapeutic strategies that can effectively manage hemodynamic instability while minimizing the risks of fluid overload. In adult patients, the early use of vasopressors has been recommended to restore perfusion in patients with septic shock, compared to repeated fluid loading. However, previous research on the use of norepinephrine and the preload status of the pediatric population is still limited. In addition, the use of fluid resuscitation does not always exhibit the desirable response, which is the increase of blood pressure. This is because the blood pressure depends not only on the stroke volume but also the vascular resistance. Consequently, predicting blood pressure elevation after fluid resuscitation remains challenging. Based on previous research, arterial elastance has the potential to predict the increase of blood pressure in response to fluid administration. Thus, this study aimed to investigate the effects of early administration of fluid resuscitation combined with norepinephrine in pediatric septic shock patients and evaluate the useof arterial elastance as a predictor of blood pressure response following fluid resuscitation. Finally, this study will also evaluate the parameters such as stroke volume index, cardiac index, lactate clearance , arterial elastance in pediatric patients with septic shock who were resuscitated using the hemodynamic support guidelines according to the Surviving Sepsis Campaign protocols.

DETAILED DESCRIPTION:
The complexity of pediatric septic shock arise from its varied pathophysiology, which includes systemic inflammation, cardiovascular collapse, and multiple organ dysfunction. Current standard treatments, which primarily focused on fluid resuscitation, had exhibited several problems. Excessive fluid resuscitation has been associated with complications such as fluid overload, which may cause conditions such as pulmonary edema and organ dysfunction, leading to worsened outcomes. This emphasizes the need for alternative therapeutic strategies that can effectively manage hemodynamic instability while minimizing the risks of fluid overload. In adult patients, the early use of vasopressors has been recommended to restore perfusion in patients with septic shock, compared to repeated fluid loading. However, previous research on the use of norepinephrine and the preload status of the pediatric population is still limited. In addition, the use of fluid resuscitation does not always exhibit the desirable response, which is the increase of blood pressure. This is because the blood pressure depends not only on the stroke volumebut also the vascular resistance. Consequently, predicting blood pressure elevation after fluid resuscitation remains challenging. Based on previous research, arterial elastance has the potential to predict the increase of blood pressure in response to fluid administration. Thus, this study aimed to investigate the effects of early administration of fluid resuscitation combined with norepinephrine in pediatric septic shock patients and evaluate the use of arterial elastance as a predictor of blood pressure response following fluid resuscitation. Finally, this study will also evaluate the parameters such as stroke volume index, cardiac index, lactate clearance , arterial elastance in pediatric patients with septic shock who were resuscitated using the hemodynamic support guidelines according to the Surviving Sepsis Campaign protocols.

Research Objectives

1. Evaluate the changes in preload between the pediatric septic shock patients receiving fluid loading with early administration of norepinephrine compared to those who only receive fluid loading.
2. Evaluate the changes in stroke volume index, cardiac index, and mean arterial pressure between the pediatric before and after treatment in both groups.
3. Evaluate the changes in lactate clearance before and after treatment in both groups.
4. Assess the sensitivity and specificity of arterial elastance as a predictor of blood pressure response in patients receiving fluid resuscitation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 3 months to 18 years with critical condition
2. Suspected or confirmed infection, indicated by fever accompanied by signs of shock:

   1. Mean arterial pressure 5th percentile, or
   2. Systolic pressure ≤ 5th percentile, or
   3. Diastolic pressure ≤ 5th percentile, or
   4. Wide pulse pressure (diastolic pressure < half of systolic pressure), or
   5. Tachycardia accompanied by one or more of the following signs: Altered mental status, capillary refill time > 2 seconds, temperature difference between extremities and core body, weaker peripheral arterial pulsation compared to the central pulsation, bounding pulse, mottled skin.

Exclusion Criteria:

1. Contraindication of fluid loading (signs of fluid overload)
2. Burn injury, massive bleeding, dengue hemorrhagic fever.
3. Cardiogenic shock.
4. Deep anesthesia.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
stroke volume index | evaluate one hour after intervention
  Evaluate the changes in stroke volume index using Ultrasonic Cardiac Output Monitor (USCOM), in units ml/m2, between the pediatric septic shock patients receiving fluid loading with early norepinephrine compared to those who only receive fluid loading
cardiac index | evaluate one hour after intervention
  Evaluate the changes in cardiac index Ultrasonic Cardiac Output Monitor (USCOM), in units L/m2/minute,between the pediatric septic shock patients receiving fluid loading with early norepinephrine compared to those who only receive fluid loading
Lactate | evaluate one hour after intervention
  Lactate clearance is defined as the change in lactate levels between two time points and is expressed as a 10-20% reduction in lactate per hour or a reduction of at least 10% within 6 hours during initial resuscitation

SECONDARY OUTCOMES:
arterial elastance | evaluate one hour after intervention
  Arterial elastance is obtained using the formula: (0.9 x systolic blood pressure)/stroke volume or mean arterial pressure/stroke volume
pulmonary edema | evaluate one hour after intervention
  pulmonary edema shown by B-line using lung ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Sugimoto M, Manabe H, Nakau K, Furuya A, Okushima K, Fujiyasu H, Kakuya F, Goh K, Fujieda K, Kajino H. The role of N-terminal pro-B-type natriuretic peptide in the diagnosis of congestive heart failure in children. - Correlation with the heart failure score and comparison with B-type natriuretic peptide -. Circ J. 2010 May;74(5):998-1005. doi: 10.1253/circj.cj-09-0535. Epub 2010 Apr 6. PMID 20378998
- [Result] Maitland K, Kiguli S, Opoka RO, Engoru C, Olupot-Olupot P, Akech SO, Nyeko R, Mtove G, Reyburn H, Lang T, Brent B, Evans JA, Tibenderana JK, Crawley J, Russell EC, Levin M, Babiker AG, Gibb DM; FEAST Trial Group. Mortality after fluid bolus in African children with severe infection. N Engl J Med. 2011 Jun 30;364(26):2483-95. doi: 10.1056/NEJMoa1101549. Epub 2011 May 26. PMID 21615299
- [Result] Macdonald S, Peake SL, Corfield AR, Delaney A. Fluids or vasopressors for the initial resuscitation of septic shock. Front Med (Lausanne). 2022 Nov 24;9:1069782. doi: 10.3389/fmed.2022.1069782. eCollection 2022. PMID 36507525
- [Result] Garcia MI, Romero MG, Cano AG, Aya HD, Rhodes A, Grounds RM, Cecconi M. Dynamic arterial elastance as a predictor of arterial pressure response to fluid administration: a validation study. Crit Care. 2014 Nov 19;18(6):626. doi: 10.1186/s13054-014-0626-6. PMID 25407570
- [Result] Choudhary R, Sitaraman S, Choudhary A. Lactate clearance as the predictor of outcome in pediatric septic shock. J Emerg Trauma Shock. 2017 Apr-Jun;10(2):55-59. doi: 10.4103/JETS.JETS_103_16. PMID 28367008